CLINICAL TRIAL: NCT06482827
Title: Effects of Repetitive Transcranial Magnetic Stimulation on Neuropathy in Diabetic Neuropathy: A Pilot Study
Brief Title: Treatment for Diabetic Neuropathy Using Repetitive Transcranial Magnetic Stimulation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Aimee Nelson, Proffessor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17797
Record Dates: First submitted 2024-06-26; First posted 2024-07-01 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Diabetic Neuropathies
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Sham) (Sham Comparator): Participants in group A will take part in 4 weeks of treatment with 5 sessions per week. Each session will involve sham repetitive transcranial magnetic stimulation (rTMS). Sham rTMS will be delivered at 10 Hz, 2004 pulses targeting the leg representation of the primary motor cortex. Participants will hear and experience the clicking but will not be provided with any stimulation. Sham rTMS will take approximately 11.5 minutes.
  Interventions: Device: Sham Repetitive transcranial magnetic stimulation
- Group B (Active) (Active Comparator): Participants in group B will take part in 4 weeks of treatment with 5 sessions per week. Each session will involve real repetitive transcranial magnetic stimulation (rTMS). rTMS will be delivered at 10 Hz, 2004 pulses targeting the leg representation of the primary motor cortex. rTMS will take approximately 11.5 minutes.
  Interventions: Device: Repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: Sham Repetitive transcranial magnetic stimulation — Sham repetitive transcranial magnetic stimulation (rTMS) is a non-invasive, non-painful procedure. The abductor pollicis brevis (APB) muscle of the left motor cortex will be targeted using neuronavigation software. During the sham, participants will hear and experience the clicking from the device but will not be provided with any stimulation. The delivery of sham rTMS requires ~ 11.5 minutes in total.
  Arms: Group A (Sham)
Device: Repetitive transcranial magnetic stimulation — Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive, non-painful procedure used to relieve chronic pain and promote short-term changes. The abductor pollicis brevis (APB) muscle of the left motor cortex will be targeted using neuronavigation software. 2004 pulses will be delivered at 10 Hz stimulation. Stimulation will be delivered at 80% of the resting motor threshold obtained from the right APB muscle. The delivery of rTMS requires ~ 11.5 minutes in total.
  Other Names: rTMS, Repetitive TMS
  Arms: Group B (Active)

SUMMARY:
The aim of this study is to determine whether a 4-week treatment of repetitive transcranial magnetic stimulation (rTMS) can alleviate the symptoms of neuropathy in individuals with diabetic neuropathy. The study will involve using questionnaires, nerve assessments, sensory tests, blood flow measurements, and blood tests to monitor any changes in symptoms after the rTMS intervention.

DETAILED DESCRIPTION:
Diabetic neuropathy (DN) is one of the most common complications of diabetes, occurring in ~50% of patients. DN results from damage to the peripheral and autonomic nervous systems. Due to the damage to small peripheral nerve fibers, patients often do not properly perceive local traumas because of the absence of pain perception and vibration perception. The upper and lower limbs are the most commonly affected areas among individuals with DN, putting patients at a higher risk of developing skin ulcerations and undergoing amputations. DN is characterized by various symptoms including numbness, loss of sensation, tingling, weakness, pain, unsteadiness, loss of vibration sense and abnormal temperature (often cold). DN is associated with decreased quality of life, depression, sleep disturbance and anxiety. It is currently managed by the control of blood glucose levels, medications to relieve pain and symptoms, physical therapy and lifestyle modifications. The global prevalence of DN is increasing, leading to a high incidence of lower limp amputations in the DN population, which accounts for approximately 70% of non-traumatic amputations worldwide. DN is also correlated with increased risk of cardiovascular disease and leads to an increase in mortality of diabetic patients. Therefore, it is crucial to find new ways to improve neuropathy in patients living with DN.

A novel approach to treating neuropathy is through the induction of neuroplasticity. Neuroplasticity refers to the ability of the brain to change, either through structural reorganization or functional changes in brain activation. Neuroplasticity can be induced non-invasively with a form of brain stimulation known as repetitive Transcranial Magnetic Stimulation (rTMS). rTMS involves an electromagnetic coil placed against the scalp that generates magnetic pulses to induce electric fields in the brain. By delivering these electric fields in rapid succession and at low intensity, functional changes in the brain (i.e. neuroplasticity) can be evoked. rTMS can be used to treat neurodegeneration, blood flow change, autonomic nervous disorders, depression, and vascular endothelial injury. rTMS can produce inhibitory or excitatory stimulation of the cerebral cortex or specific areas, leading to remodeling of the nervous system. This makes it a promising application for promoting nerve regeneration, neuroprotection, and localization of injuries. DN is closely related to cardiovascular disease as DN damages the autonomic nervous system (ANS), which controls heart rate (HR) and blood pressure (BP). With rTMS, this damage in ANS, specifically, HR and BP, can be improved. Inhibitory stimulation can lower HR while excitatory stimulation can enhance heart rate variability. Both inhibitory and excitatory stimulation can lower BP. Thus, the use of rTMS can improve a variety of functions that could prevent further complications and possibly improve neuropathy, as well.

Inflammation is a crucial factor in the progression of DN, as it involves an increase in chemokine production, inflammatory cell infiltration in the kidney, tissue damage, and production of pro-inflammatory cytokines. Infiltration of inflammatory cells into the kidney can lead to diabetic kidney disease, which is the most prevalent cause of terminal renal failure globally with suboptimal treatment options. Due to the close link between DN and inflammation, reducing inflammation has been suggested as a possible therapeutic option for this population. Additionally, diabetic wounds and inflammation are also associated, therefore controlling inflammation may improve wound management and healing rates. Researchers have recently discovered that rTMS can impact the levels of inflammatory markers (such as IL-1B, IL-6, IL-10, TNF-α, TGF-β, CRP, SP, and BDNF) in other conditions such as depression, post-stroke, and Alzheimer's. The study by Zhao et al. investigated the effects of 20 sessions of rTMS intervention on 29 individuals diagnosed with refractory depression. Significant increases in serum BDNF levels and decreases in IL-1β and TNF-α levels were noted after one week of intervention, compared to healthy individuals, and this trend continued over the 4-week stimulation period. However, there was no change noted in the sham group. Cha et al. conducted a post-stroke study measuring the effects of 10 sessions of rTMS intervention on 10 individuals with post-stroke cognitive impairment. Following the intervention, levels of IL-1β, IL-6, TNF-α, and TGF-β mRNA decreased. Velioglu et al. explored the effects of 10 sessions of rTMS intervention on 15 individuals with Alzheimer's Disease. An increase in BDNF levels was noted following the conclusion of the intervention. Although no studies have been done in the DN population, the use of rTMS to examine changes in these levels is promising.

The goal of the proposed research is to investigate the use of rTMS to improve the symptoms of neuropathy in patients living with diabetic neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of diabetic neuropathy

Exclusion Criteria:

* Contraindications to transcranial magnetic stimulation
* Known psychological diagnosis affecting comprehension
* Inability to participate in the study

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Modified Toronto Clinical Neuropathy Score | Immediately before intervention, immediately following intervention, 4 weeks after intervention
  Will be used to assess the presence and severity of diabetic neuropathy ('yes' or 'no')
PROMIS-29 v2.0 Profile | Immediately before intervention, immediately following intervention, 4 weeks after intervention
  Using numerical rating (0 to 5) to assess seven health domains including physical function, anxiety, depression, fatigue, sleep disturbances, ability to participate in social roles and activities, and pain interference. Each category consists of 4 questions. Also uses a numerical rating to asses pain intensity (0-10).
Patient Perceived Global Index of Change (PGIC) | Immediately following intervention, 4 weeks after intervention
  1-7 Likert Scale: Patients rate their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse
Pain catastrophizing scale-EN-SF | Immediately before intervention, immediately following intervention, 4 weeks after intervention
  Will be used to assess the patients feeling and emotion related to their pain experience

SECONDARY OUTCOMES:
Change in quantitative sensory testing | Immediately before intervention, immediately following intervention, 4 weeks after intervention
  Will be used in this study to assess somatosensory function to determine underlying pain mechanisms for pain phenotypes. QST will be used to measure detection thresholds for cold, warm, vibration, and mechanical stimuli. Pain thresholds will be assessed for cold, heat, mechanical, and pressure stimuli. In addition, allodynia will be measured.
Change in nerve conduction assessments | Immediately before intervention, immediately following intervention
  Non-invasive peripheral nerve stimulation will be delivered using surface bar electrodes placed over the tibial nerve at the popliteal fossa and the medial malleolus. Compound muscle action potential will be recorded with surface electromyography over soleus, gastrocnemius, and abductor hallucis. These measures will be obtained from both lower limbs.
Change in blood flow | Immediately before intervention, immediately following intervention
  Will use color Doppler ultrasound to measure hemodynamic characteristics in diabetic neuropathy. Six major arteries that are responsible for supplying blood to the foot sole will be evaluated including the first common plantar artery, second common plantar artery, third common plantar artery, fourth common plantar artery, posterior tibial artery, and fibular side of the first plantar toe proper artery.
Changes in wound | Immediately before intervention, immediately following intervention
  Will use the app called Swift Skin and Wound to track the changes in wound size over the course of the study
Change in inflammation markers (IL-1B, IL-6, IL-10, TNF-α, TGF-β, CRP, SP, and BDNF) | Immediately before intervention, immediately following intervention
  10 mL of blood will be collected to assess the changes in the levels of inflammatory markers (IL-1B, IL-6, IL-10, TNF-α, TGF-β, CRP, SP, and BDNF)

CONTACTS AND LOCATIONS:
Overall Officials: Aimee Nelson, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- See also: Ader, D. N. (2007). Developing the Patient-Reported Outcomes Measurement Information System (PROMIS). Medical Care, 45(5), S1. — https://doi.org/10.1097/01.mlr.0000260537.45076.74
- See also: Bondar, A. C., & Popa, A. R. (2018). Diabetic Neuropathy Prevalence and Its Associated Risk Factors in Two Representative Groups of Type 1 and Type 2 Diabetes Mellitus Patients from Bihor County. Mædica, 13(3), 229-234. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6290177/
- See also: Callaghan, B., Kerber, K., Langa, K. M., Banerjee, M., Rodgers, A., McCammon, R., Burke, J., & Feldman, E. (2015). Longitudinal patient-oriented outcomes in neuropathy. Neurology, 85(1), 71-79. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4501944/
- See also: Cha, B. et al. (2022). Therapeutic Effect of Repetitive Transcranial Magnetic Stimulation for Post-stroke Vascular Cognitive Impairment: A Prospective Pilot Study. Frontiers in Neurology, 13. — https://doi.org/10.3389/fneur.2022.813597
- See also: Defrin, R et al. (2007). The effect of a series of repetitive transcranial magnetic stimulations of the motor cortex on central pain after spinal cord injury. Archives of Physical Medicine and Rehabilitation, 88(12), 1574-1580. — https://doi.org/10.1016/j.apmr.2007.07.025
- See also: Duran-Salgado, M. B., & Rubio-Guerra, A. F. (2014). Diabetic nephropathy and inflammation. World Journal of Diabetes, 5(3), 393-398. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4058744/
- See also: Feldman, E. L., Callaghan, B. C., Pop-Busui, R., Zochodne, D. W., Wright, D. E., Bennett, D. L., Bril, V., Russell, J. W., & Viswanathan, V. (2019). Diabetic neuropathy. Nature Reviews. Disease Primers, 5(1), 42. — https://doi.org/10.1038/s41572-019-0097-9
- See also: Ferguson, L., & Scheman, J. (2009). Patient global impression of change scores within the context of a chronic pain rehabilitation program. The Journal of Pain, 10(4), S73. — https://doi.org/10.1016/j.jpain.2009.01.258
- See also: Foglia, S. D. et al. (2022). Case report: The feasibility of rTMS with intrathecal baclofen pump for the treatment of unresolved neuropathic pain following spinal cord injury. Frontiers in Rehabilitation Sciences, 3, 893014. — https://doi.org/10.3389/fresc.2022.893014
- See also: Hallett, M. (2007). Transcranial Magnetic Stimulation: A Primer. Neuron, 55(2), 187-199 — https://doi.org/10.1016/j.neuron.2007.06.026
- See also: Juster-Switlyk, K., & Smith, A. G. (2016). Updates in diabetic peripheral neuropathy. F1000Research, 5, F1000 Faculty Rev-738. — https://doi.org/10.12688/f1000research.7898.1
- See also: Kang, B. S., Shin, H. I., & Bang, M. S. (2009). Effect of repetitive transcranial magnetic stimulation over the hand motor cortical area on central pain after spinal cord injury. Archives of Physical Medicine and Rehabilitation, 90(10), 1766-1771. — https://doi.org/10.1016/j.apmr.2009.04.008
- See also: Lee, H., Lee, J. H., Hwang, M.-H., & Kang, N. (2023). Repetitive transcranial magnetic stimulation improves cardiovascular autonomic nervous system control: A meta-analysis. Journal of Affective Disorders, 339, 443-453. — https://doi.org/10.1016/j.jad.2023.07.039
- See also: Lim, A. K. H., & Tesch, G. H. (2012). Inflammation in Diabetic Nephropathy. Mediators of Inflammation, 2012(1), 146154. — https://pubmed.ncbi.nlm.nih.gov/22969168/
- See also: Pop-Busui, R., Ang, L., Holmes, C., Gallagher, K., & Feldman, E. L. (2016). Inflammation as a Therapeutic Target for Diabetic Neuropathies. Current Diabetes Reports, 16(3), 29. — https://doi.org/10.1007/s11892-016-0727-5
- See also: Sieberg, C. B., Taras, C., Gomaa, A., Nickerson, C., Wong, C., Ward, C., Baskozos, G., Bennett, D. L. H., Ramirez, J. D., Themistocleous, A. C., Rice, A. S. C., Shillo, P. R., Tesfaye, S., Edwards, R. R., Andrews, N. A., Berde, C., & Costigan, M. (2018). — https://doi.org/10.1097/PR9.0000000000000651
- See also: Vinik, A. I., Erbas, T., & Casellini, C. M. (2013). Diabetic cardiac autonomic neuropathy, inflammation and cardiovascular disease. Journal of Diabetes Investigation, 4(1), 4-18. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3580884/
- See also: Xu, X., & Xu, D.-S. (2021). Prospects for the application of transcranial magnetic stimulation in diabetic neuropathy. Neural Regeneration Research, 16, 955. — https://doi.org/10.4103/1673-5374.297062
- See also: Yang, S., Kwak, S. G., Choi, G.-S., & Chang, M. C. (2022). Short-term Effect of Repetitive Transcranial Magnetic Stimulation on Diabetic Peripheral Neuropathic Pain. Pain Physician, 25(2), E203-E209. — https://pubmed.ncbi.nlm.nih.gov/35322973/